CLINICAL TRIAL: NCT03129984
Title: A Mandibular Movement Test as a Screening Tool for Polysomnography Candidates Among Patients With Sleep Apnea: a Retrospective Feasibility Study
Brief Title: Mandibular Movement Test as a Screening Tool for Polysomnography Candidates
Acronym: dépist-By
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: nomics s.a. (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0148
Record Dates: First submitted 2017-04-21; First posted 2017-04-26 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-04

CONDITIONS: Sleep Apnea Syndromes
Keywords: mandibular movements
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: The study population is comprised of all patients included in the Brizzy register, Belgium.
  Interventions: Device: Mandibular movement tracking

INTERVENTIONS:
Device: Mandibular movement tracking — Patients wore the Brizzy device while sleeping. Mandibular movements (A mid-sagittal mandibular movement magnetic sensor measured the distance in mm between two parallel, coupled, resonant circuits placed on the forehead and chin.) were tracked during sleep.
  Other Names: Brizzy (Nomics, Liege, Belgium)

SUMMARY:
The primary objective of this study is to determine the technical failure and inconclusive test rates when using the Brizzy device for mandibular movement tracking.

ELIGIBILITY:
Inclusion Criteria:

* Patient included in the Brizzy register
* Mandibular movement test prescribed by practitioner
* Patient performed a mandibular movement test (ambulatory setting) using a magnetic sensor (Brizzy, Nomics, Liege, Belgium)

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is re-evaluating data provided by the Brizzy register in Belgium.
Sampling Method: Probability Sample
Enrollment: 4231 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The exploitable data rate | Day 0 (retrospective cross-sectional study)
  The number of usable tests / the number of tests performed.

SECONDARY OUTCOMES:
Respiratory disturbance index based on mandibular movements | Day 0 (retrospective cross-sectional study)
  Respiratory disturbance index based on mandibular movements (Brizzy, Nomics, Liege, Belgium)
Minimal estimated total sleep time | Day 0 (retrospective cross-sectional study)
  Minimal estimated total sleep time
ODI | Day 0 (retrospective cross-sectional study)
  The oxygen desaturation index (ODI) from oximetry.
Type of prescriber (qualitative) | Day 0 (retrospective cross-sectional study)
  Was the prescriber a (choose one from among the following):
  * cardiologist,
  * general practitioner
  * otorhinolaryngologist
  * pneumologist
  * orthodontist
  * other
Identification of reasons why a given test was unusable | Day 0 (retrospective cross-sectional study)
age | Day 0 (retrospective cross-sectional study)
  age in years

CONTACTS AND LOCATIONS:
Overall Officials: Dany Jaffuel, MD, PhD, Study Director — University Hospitals of Montpellier

REFERENCES:
- [Derived] Rotty MC, Mallet JP, Borel JC, Suehs CM, Bourdin A, Molinari N, Jaffuel D. The feasibility of a mandibular movement test as a screening tool for polysomnography candidates. Eur Respir J. 2017 Nov 30;50(5):1701076. doi: 10.1183/13993003.01076-2017. Print 2017 Nov. No abstract available. PMID 29191954